CLINICAL TRIAL: NCT03563079
Title: Effects of Instrument-assisted Soft Tissue Mobilization (IASTM) on Pain and Disability in Individuals With Non-specific Chronic Neck Pain: A Randomized Clinical Trial
Brief Title: Effects of Instrument-assisted Soft Tissue Mobilization (IASTM) on Pain and Disability in Individuals With Non-specific Chronic Neck Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Francisco Xavier de Araujo, Pt, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAraujo
Record Dates: First submitted 2018-05-25; First posted 2018-06-20 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Neck Pain; Myofascial Pain Syndrome
Keywords: Handling, Musculoskeletal; Tissue, Subcutaneous; Myofascial Release; Instrument-Mobilized Soft Tissue Mobilization
MeSH Terms: conditions — Neck Pain; Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Participants selected to participate in this research will be randomly drawn and randomly allocated using sealed opaque envelopes, and therefore included randomly in one of the two groups present in this study. A collaborative researcher blind to the groups will be assigned to conduct the pre- and post-intervention evaluation process of all individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental): The treatment will be performed using two pieces of Instrument Assisted Soft Tissue Mobilization (IASTM) stainless steel in the neck, bilaterally, which comprise the following muscles: Upper Trapezius, Splenius, scalenes and Sternocleidomastoid. An established time of 3 minutes will be used in each region, using an angle of 30 to 60º with the instrument. As it is observed, through the instrument, regions of greater adhesion, the researcher will use most of this time to release this condition.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization
- group control (Active Comparator): Treatment will be performed using manual Myofascial Release techniques. Release the upper Trapezius muscle bilaterally, sliding using roller with the dorsum of the fingers and ending with myofascial release. Sternocleidomastoid, sliding using roller with the dorsum of the fingers, ending with myofascial release. Afterwards the release of the scalenes muscles will be performed, with the fingers sliding and ending with the myofascial release. Soon afterwards techniques will be performed for the Splenius muscles, using finger slips and ending with posterior cervicothoracic release. The same time of 3 min will be used for the treatment bilaterally in each region.
  Interventions: Other: Manual Myofascial Release

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization — Soft Tissue Mobilization
  Other Names: IASTM
  Arms: trial group
Other: Manual Myofascial Release — Myofascial Release Technique
  Arms: group control

SUMMARY:
INTRODUCTION: Cervical pain is a very common clinical condition in the world population, and can affect 70% of people at some point in life. Many of these conditions arise from musculoskeletal disorders, which may be caused by myofascial dysfunctions. Instrument-assisted soft tissue mobilization (IASTM) may be an important therapeutic tool as a means of treatment under these conditions. PURPOSE: To verify the effect of instrument-assisted soft tissue mobilization (IASTM) on pain, disability and range of motion (ROM) in individuals with non-specific chronic neck pain. DESIGN: Randomized Clinical Trial. METHODS: The sample will consist of 46 volunteers with non-specific chronic neck pain of both sexes, aged between 18 and 60 years, who presented pain for at least 12 weeks, without irradiation to the upper limbs distally to the shoulders. Of these, those that are not excluded, will be allocated randomly in one of the two groups present: Experimental Group (GE) - IASTM in the neck and Control Group (CG) - Manual myofascial release in the neck region. A blinded evaluator will be assigned to conduct the evaluation process for both groups. DESPECTS: The outcomes will be neck pain, neck disability and range of motion of the neck.

DETAILED DESCRIPTION:
* To verify the effect of instrument-assisted soft tissue mobilization (IASTM) on pain, disability and ROM in individuals with non-specific chronic neck pain.
* Characterization of individuals with chronic nonspecific neck pain. To describe and compare, at the pre-intervention, post-intervention moments in a 3-week follow-up period, the intensity of neck pain using the numerical pain scale (NPS); the self - perception of disability using the Neck Disability Index (NDI) and range of motion (ROM) of the neck - flexion, extension, rotations and right and left slopes through a pendulum flexometer.
* Randomized unicentric clinical trial of longitudinal cut according to the standardization proposed by the Consolidated Standards of Reporting Trials - CONSORT statement
* The sample will be composed of 46 volunteers with chronic nonspecific neck pain.
* The subjects will be recruited through digital ads in the main social networks, as well as coming from the Physiotherapy service in a clinic in the city of Viamão / RS. An online form will be completed by the interested parties, which will include the eligibility criteria for participation in the study. Only the subjects that follow the criteria will be allocated to carry out the study.

ELIGIBILITY:
Inclusion Criteria:

* people presenting as main complaint chronic neck pain, manifested for at least twelve weeks, without irradiation to the upper limbs distally to the shoulders.
* presenting scales scores (NSP) above 3 and NDI above 30%.

Exclusion Criteria:

* Individuals who are positive in the Spurling test, indicating Cervical Radiculopathy,
* Some severe clinical condition (such as fracture, neoplasia or systemic diseases); --
* history of previous surgery in the neck or thoracic spine;
* injury of whiplash trauma in the six months prior to evaluation;
* diagnosis of cervical stenosis;
* diagnosis of myelopathy;
* pregnancy;
* signs and symptoms of moderate to severe temporomandibular dysfunction,
* neck hematoma,
* neck scarring,
* severe osteoporosis,
* open lesions or recent neck fractures,
* generalized infections,
* coagulation disorders,
* acute inflammatory conditions,
* fever.
* Also excluded are patients who have undergone physical therapy or massage up to one month prior to the evaluation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-04-20 (Estimated); Study Completion 2019-05-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pain | assessment at baseline and its change in 1-week and 3-month follow-up
  the numerical scale of pain will be used. The Numerical Scale consists of a ruler divided into equal parts, numbered successively from 0 to 10. The study participant is meant to make the equivalence between the intensity of his pain and a numerical classification, where 0 corresponds to the classification "No Pain" and 10 to the classification "Maximum Pain" (pain of maximum intensity imaginable), that is, the higher the number the worse the score.
Disability of the neck | assessment at baseline and its change in 1-week and 3-month follow-up
  Neck disability index. The Neck Disability Index is used to assess the functional capacity of the neck. Is composed of 10 questions regarding activities and pain. Items are organized by type of activity and followed by six different statements expressing progressive functional capacity levels. The NDI score consists of the sum of the points, from 0 to 5 of each of the 10 questions, totaling a maximum of 50 points. O value can be expressed as a percentage, on a scale of 0% (no disability) to 100% (complete disability). The score total is divided by the number of questions answered multiplied by number 5. The higher the score, the greater the patient's disability.
Range of motion | assessment at baseline and its change in 1-week and 3-month follow-up
  For measurement, an angular flexometer

SECONDARY OUTCOMES:
characterization of the sample | baseline
  quiz

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Federal university of health sciences of porto alegre, Porto Alegre, Rio Grande do Sul
  - Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No